CLINICAL TRIAL: NCT07263646
Title: The Effect of Balance-focused Exercise Programme in Enhancing the Solus-muscle Activation During Gait Initiation for People With Parkinson Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Kuwait (Other Government)
Responsible Party: Principal Investigator, Esraa Aldayil, chief of physiotherapy, Ministry of Health, Kuwait
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2824/2025
Record Dates: First submitted 2025-07-15; First posted 2025-12-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease; Gait Disorders; Gait Balance
Keywords: gait initiation; Parkinson disease; rehabilitation; balance-focus exercise
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: parallel group prospective (10 weeks) randomised single-blinded controlled trial
Who Masked: Outcomes Assessor
Masking Description: the outcomes assessor will not be aware of the group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): Control Group: Conventional Physiotherapy - Participants will receive standard physiotherapy interventions targeting gait and motor symptoms.
  Conventional Physiotherapy will include:
  * Balance and Postural Training, (e.g. bridging and rolling exercise),
  * Flexibility and Range of Motion (e.g. upper limb exercise include shoulder, elbow and wrist movements, lower limb exercise including hip, knee and ankle movement)
  * Strength Training focus on anti-gravity muscles (e.g. squatting, body-weight strengthening exercise)
  * Functional Mobility Training (e.g. Sit-to-stand practice and stairs training
  * gait training (e.g. Practice heel-to-toe walking, emphasize large, exaggerated steps, use visual cues and auditory cues, turn training: wide arc turning to avoid freezing, treadmill walking with therapist supervision)
  * home program.
- intervention (treatment ) group (Experimental): Participants will receive comprehensive balance-focused exercise programme integrated into conventional physiotherapy. The participants will be engaged in supervised sessions (by physiotherapists) of interactive balanced exercises focusing on improving balance, cognition, and coordination. The comprehensive balance-focused exercise programme will consist of motor tasks using interactive balance device to facilitate postural stability and weight-shifting control.
  Interventions: Other: balance-focus exercise programe

INTERVENTIONS:
Other: balance-focus exercise programe — participants in the experimental group will receive balance-focused exercise programe integrated into conventional physiotherapy programe provided to people with parkinson.
  Arms: intervention (treatment ) group

SUMMARY:
Gait initiation (GI) is a crucial component of walking that requires a balanced muscle activity and postural stability. GI could be challenging for people with neurological condition such as people with Parkinson (PWP), where GI is usually impaired. The purpose of this study is determining effectiveness of comprehensive, balanced-focused exercise programme in controlling the activation of Solus-muscle in people with Parkinson disease. We hypothesise that balance-focus exercise programe could improve Solus-muscle activation during GI.

study type: this is a parallel group prospective (10 weeks) randomised single-blinded controlled trial conduct in Kuwait.

Participant: People with Parkinson, who met the inclusion criteria.

DETAILED DESCRIPTION:
Parkinson's Disease (PD), a neurodegenerative disorder characterised by motor dysfunction . The basal ganglia play a significant role in regulating muscle excitation, and its dysfunction in PD leads to abnormal activation patterns in muscles such as the soleus, crucial for walking. This contributes to symptoms like bradykinesia, resulting in slower movement, shuffling gait, and difficulty initiating walking. Prolonged activation of the plantar flexor muscles, especially the soleus, disrupts the forward momentum needed for normal walking.

Gait initiation (GI) is a crucial component of walking that requires a balanced muscle activity and postural stability. The GI process requires a propulsive force to move the body across a distance (from a bipedal stance to repeating gait cycles) while maintaining postural stability. Thus, GI could be challenging for people with neurological condition such as people with Parkinson (PWP), where GI is usually impaired.

Any modification to the GI program could affect postural stability and the velocity of the movement and any impairment in muscle activation of the lower limb will interfere with the GI process, .

This underscores the significance of the altered muscle excitation pattern observed in PWP and its potential impact on motor control. This imbalance can contribute to the prolonged muscle activation times and differential speed changes observed in muscle activation patterns.

Bradykinesia is a slow movement during the execution of common physical activities, such as the activities of daily living (ADL). That could be because PWP tend to keep the plantar flexor muscles mainly (solus) contracted for longer time. This prolonged muscle activity interferes with the gravity-assisted forward rotation of the body resulting adverse affects on the timing of subsequent events during gait initiation.

Therefore, therapies aimed at restoring the balance during GI may help improve motor control and balance in individuals, thus improve GI speed with Parkinson's disease.

Balance-focused rehabilitation strategies, including interactive exercises, are promising in addressing delays in GI. Several previous studies explored the effect of balance exercise of the GI in patients with Parkinson. For example, in a systematic exploration of cueing therapy's impact on gait and balance in individuals with Parkinson's disease, revealed its efficacy. This approach, the cueing therapy was highlighted as a promising intervention for addressing gait and balance challenges in Parkinson's disease. Another significant approach for functional rehabilitation is the utilization of balance boards, as underscored by. Investigating the effectiveness of a Wii Fit™-based balance board exercise program in the elderly population. Consequently, Mhatre et al. concluded that the Wii Fit™ balance board exercise program represents a valuable tool for augmenting balance and mitigating fall risk among older adults. In the context of functional rehabilitation, these interventions, particularly cueing therapy and balance board exercises, signify promising avenues for improving motor function and addressing challenges associated with gait and balance. Consideration of these therapeutic approaches is crucial for devising comprehensive and effective rehabilitation strategies tailored to the unique needs of individuals undergoing functional rehabilitation.

However, there is a need for further research to explore effective rehabilitation strategies tailored to different disease severity levels. To improve the maintenance and rehabilitation of community walking ability in PWP, there is a need to understand the details of the kinematics, as well as the muscle activation characteristics during while GI.

ELIGIBILITY:
Inclusion Criteria:

* participants diagnosed by their neurologist with Parkinson's disease (moderate to severe stage)
* stable on anti-Parkinson's drugs
* able to walk independently without a frame or walking stick.
* Able to walk for more than 10 mins unaided
* without cognitive disability (Able to follow simple instructions and communicate, orally),
* have good vision (with or without corrective aids)

Exclusion Criteria:

* are pregnant
* cardiac problems exacerbated by exercise
* currently complaining of joint or muscle problems that affect walking ability
* known to have neurological conditions (other than Parkinson) that affect walking ability
* uncorrected hearing or vision problems
* history of severe motion sickness
* history of vestibular or balance problems
* an active skin condition that could be irritated by contact with sticky tape.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2027-12-22 (Estimated); Study Completion 2028-12-22 (Estimated)

PRIMARY OUTCOMES:
weight | baseline
  weight of the person in KG
height | baseline
  the height of the person in CM
gait analysis | baseline
  • Three-dimensional motion analysis:Motion capture units will track the movement of reflective markers placed on the skin/clothing of participants.
Gait Analysis | 6 weeks
  Three-dimensional motion analysis: Motion capture units will track the movement of reflective markers placed on the skin/clothing of participants.
gait analysis | 10 weeks
  Three-dimensional motion analysis: Motion capture units will track the movement of reflective markers placed on the skin/clothing of participants.
• electromyography (EMG) | baseline
  Electric activity of the muscles using the wireless EMG measurement system. The system will track the activity of solus muscle (left and right).
electromyography EMG | 6 weeks
  Electric activity of the muscles using the wireless EMG measurement system. The system will track the activity of solus muscle (left and right).
electromyography EMG | 10 weeks
  Electric activity of the muscles using the wireless EMG measurement system. The system will track the activity of solus muscle (left and right).

SECONDARY OUTCOMES:
Parkinson severity scale (PDQ-39) | baseline
  To evaluate the impact of Parkinson's disease on different dimensions of a patient's life and monitor changes over time.
Parkinson severity scale PDQ-39 | 6 weeks
  To evaluate the impact of Parkinson's disease on different dimensions of a patient's life and monitor changes over time.
Parkinson severity scale PDQ-39 | 10 weeks
  To evaluate the impact of Parkinson's disease on different dimensions of a patient's life and monitor changes over time.
Timed Up and Go test (TUG) | baseline
  widely used clinical test to assess a person's mobility, balance, walking ability, and fall risk. It is especially useful in older adults and individuals with neurological or musculoskeletal impairment
Timed Up and Go test TUG | 6 weeks
  widely used clinical test to assess a person's mobility, balance, walking ability, and fall risk. It is especially useful in older adults and individuals with neurological or musculoskeletal impairment
time up and go TUG | 10 weeks
  widely used clinical test to assess a person's mobility, balance, walking ability, and fall risk. It is especially useful in older adults and individuals with neurological or musculoskeletal impairment
PITTSBURGH rehabilitation participation scale | 6 weeks
  a clinician-rated tool used to measure a patient's level of participation in inpatient rehabilitation therapy sessions. It focuses on observed engagement, effort, and motivation.
patient satisfaction | 6 weeks
  in response to the question how satisfied are you with the results of physiotherapy treatment? Patient will be asked tp grade their level of satisfaction on 5 points liked scale (1. Not at all satisfied, 2. Dissatisfied, 3. Natural, 4. Satisfied, 5. Very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Medicine and Rehabilitation Center, Kuwait, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided
IPD collected in this research will be owned by the ministry of health in Kuwait and restrictions apply to the availability of these data publicly. however, IPD can be available from authors upon resonable request and with permission of the ministry of health

REFERENCES:
- [Background] 1- Hassler, R. (1967) 'Private communication to O'. Hornykiewicz. Letter dated February, 9 1967. 2- Lanciego, J.L., Luquin, N. and Obeso, J.A. (2012) 'Functional neuroanatomy of the basal ganglia'. Cold Spring Harbor perspectives in medicine, 2 (12), pp. a009621. 3- Breniere, Y. and Do, M.C. (1991) 'Control of gait initiation'. Journal of motor behavior, 23 (4), pp. 235-240. 4 -Grosset, D., Fernandez, H., Grosset, K., & Okun, M. (2009). Parkinson's Disease: Clinican's Desk Reference. CRC Press. 5 Cau, N., Cimolin, V., Galli, M., Precilios, H., Tacchini, E., Santovito, C., & Capodaglio, P. (2014). Center of pressure displacements during gait initiation in individuals with obesity. Journal of neuroengineering and rehabilitation, 11(1), 1-8. 6- Mickelborough, J., Van Der Linden, M., Tallis, R., & Ennos, A. (2004). Muscle activity during gait initiation in normal elderly people. Gait & posture, 19(1), 50-57. 7- Stone, E. E., Skubic, M., & Back, J. (2014). Automated health alerts from kinect-based in-home gait measurements. 2014 36th Annual International Conference of the IEEE Engineering in Medicine and Biology Society, 8 - Lelard, T., Doutrellot, P.-L., Temfemo, A., & Ahmaidi, S. (2017). Electromyographic pattern during gait initiation differentiates yoga practitioners among physically active older subjects. Frontiers in human neuroscience, 11, 300. 9 Ivanenko, Y.P., Poppele, R.E. and Lacquaniti, F., 2004. Five basic muscle activation patterns account for muscle activity during human locomotion. The Journal of physiology, 556(1), pp.267-282. 10- Berardelli, A., Rothwell, J. C., Thompson, P. D., & Hallett, M. (2001). Pathophysiology of bradykinesia in Parkinson's disease. Brain, 124(11), 2131-2146. 11 -Sherbondy, P. S., Queale, W. S., McFarland, E. G., Mizuno, Y., & Cosgarea, A. J. (2003). Soleus and gastrocnemius muscle loading decreases anterior tibial translation in anterior cruciate ligament intact and deficient knees. The journal of knee surgery, 16(3), 152-158